#### 1 **TITLE PAGE**



VERTEX PHARMACEUTICALS INCORPORATED

# Statistical Analysis Plan (Methods)

# Protocol Number VX21-548-101 Version 5.0 (Final Analysis)

A Phase 2, Randomized, Dose-ranging, Double-blind, Placebocontrolled Study Evaluating the Efficacy and Safety of VX-548 for Acute Pain After a Bunionectomy

**Author of SAP:** 



Version: 1.0 Version Date of SAP: 03 March 2022

Vertex Pharmaceuticals Incorporated 50 Northern Avenue Boston, Massachusetts 02210-1862

#### CONFIDENTIAL

This document contains confidential information. Any use, distribution, or disclosure without the prior written consent of Vertex Pharmaceuticals Incorporated is strictly prohibited except to the extent required under applicable laws or regulations. Persons to whom the information is disclosed must be informed that the information is confidential and may not be further disclosed by them.

# 2 TABLE OF CONTENTS

| 1 | Title Page | 1 |
|---|-------------------------------------------------------------|----|
| 2 | Table of Contents | 2 |
| 3 | Modifications | 4 |
| | 3.1 Modifications to the Approved Clinical Study Protocol | 4 |
| | 3.2 Modifications to the Approved Statistical Analysis Plan | |
| 4 | Introduction | |
| 5 | Study Objectives | 5 |
| | 5.1 Primary Objective | 5 |
| | 5.2 Secondary Objectives | 5 |
| | 5.3 Other Objectives | 5 |
| 6 | Study Endpoints | |
| | 6.1 Primary Endpoint | 5 |
| | 6.1.1 Secondary Endpoints | 5 |
| | 6.1.2 Other Endpoints | 6 |
| 7 | Overall Design | 6 |
| | 7.1 Sample Size and Power | 7 |
| | 7.2 Randomization | _ |
| | 7.3 Blinding and Unblinding | |
| 8 | Analysis Sets | |
| | 8.1 All Subjects Set | |
| | 8.2 Full Analysis Set | |
| _ | 8.3 Safety Set | |
| 9 | Statistical Analysis | |
| | 9.1 General Considerations | |
| | 9.2 Background Characteristics | |
| | 9.2.1 Subject Disposition | |
| | 9.2.2 Demographics and Baseline Characteristics | |
| | 9.2.3 Medical History | |
| | 9.2.4 Prior and Concomitant Medications | |
| | 9.2.5 Study Drug Exposure and Study Drug Compliance | |
| | 9.2.6 Important Protocol Deviations | |
| | 9.3 Efficacy Analysis | |
| | 9.3.1 Analysis of Primary Endpoint | |
| | 9.3.1.1 Definition of Primary Endpoint | |
| | 9.3.1.3 Supportive Analyses | |
| | 9.3.1.4 Additional Analyses 9.3.1.5 Sensitivity Analyses | |
| | 9.3.1.6 Subgroup Analysis | |
| | 9.3.2 Analysis of Secondary Efficacy Variables | |
| | 9.3.2.1 Definition of Secondary Efficacy Variables | |
| | 9.3.2.2 Secondary Analyses | |
| | / Decinally 1 man 1000 | 17 |

| | 9.3.3 | Analysis of Other Efficacy Variables | 14 |
|---|---|---|---|
| | | 1 Definition of Other Efficacy Variables | |
| | 9.3.3 | 2 Other Analyses | 15 |
| | 9.4 Safe | ety Analysis | 16 |
| | 9.4.1 | Adverse Events | 16 |
| | 9.4.2 | Clinical Laboratory Assessments | 17 |
| | 9.4.3 | Electrocardiogram | 17 |
| | 9.4.4 | Vital Signs | 18 |
| | 9.4.5 | Physical Examination | 18 |
| 10 | Summa | ry of Interim and IDMC Analyses | 18 |
| 11 | Referen | ces | 18 |
| 12 | List of A | Appendices | 19 |
| | Appendix | A : Analysis Visit Windows for Safety and Efficacy Assessments | 19 |
| | Appendix | B : Imputation Rules for Missing Prior/Concomitant Medication Date | 21 |
| | Appendix | C : Imputation Rules for Missing AE Date and Time | 22 |
| | <b>Appendix</b> | D : Threshold Value Criteria | 23 |

#### 3 MODIFICATIONS

# 3.1 Modifications to the Approved Clinical Study Protocol

Not applicable

# 3.2 Modifications to the Approved Statistical Analysis Plan

Not applicable

#### 4 INTRODUCTION

This statistical analysis plan (SAP) for the final analysis is based on the most recent approved clinical study protocol (CSP), the most recent approved electronic case report form (eCRF), and the most recent approved eCRF completion guidelines. This SAP documents the planned statistical analysis of efficacy and safety endpoints defined in the study protocol of VX21-548-101 and provides additional details and clarifications.

The Vertex Biometrics Department will perform the final statistical analysis of the efficacy and safety data; SAS® Version 9.4 Software (SAS Institute, Cary, North Carolina, USA) or higher will be used to generate all statistical outputs (tables, figures, listings and datasets).

The SAP (Methods) will be finalized and approved before the clinical database lock for the final analysis. Any revisions to the approved SAP will be documented and approved in an amendment to the SAP prior to the clinical database lock. Any revisions made to the SAP after the clinical database lock will be documented in the clinical study report for this study.

The analysis addressing the pharmacokinetic (PK) objective of the study will be described in the Clinical Pharmacology Analysis Plan (CPAP) which will be developed separately by the Clinical Pharmacology department at Vertex Pharmaceuticals Incorporated (Vertex).

#### 5 STUDY OBJECTIVES

## 5.1 Primary Objective

• To evaluate the efficacy of VX-548 doses in treating acute pain after a bunionectomy

## 5.2 Secondary Objectives

- To evaluate the safety and tolerability of VX-548
- To evaluate the pharmacokinetics (PK) of VX-548 and its metabolite,

# 5.3 Other Objectives

• To evaluate the dose-response and exposure-response relationship

#### 6 STUDY ENDPOINTS

# 6.1 Primary Endpoint

• Time-weighted sum of the pain intensity difference (SPID) as recorded on a Numeric Pain Rating Scale (NPRS) 0 to 48 hours (SPID48) after the first dose of study drug

# 6.1.1 Secondary Endpoints

- Time-weighted SPID as recorded on an NPRS 0 to 24 hours (SPID24) after the first dose of study drug
- Proportions of subjects with  $\ge 30\%$ ,  $\ge 50\%$ , and  $\ge 70\%$  reduction in NPRS at 48 hours after the first dose of study drug
- PK parameter estimates of VX-548 and its metabolite,

• Safety and tolerability based on the incidence and type of adverse events (AEs), changes from baseline in clinically significant laboratory test results, vital signs, and ECGs

## 6.1.2 Other Endpoints

- Time to onset of "confirmed perceptible pain relief" and "meaningful pain relief" after the first dose of study drug
- Proportions of subjects with ≥30%, ≥50%, and ≥70% reduction in NPRS at 24 hours after the first dose of study drug
- Patient Global Assessment (PGA) of study drug at 48 hours after the first dose of study drug
- Percentage of subjects using rescue medication, and total rescue medication usage, 0 to 48 hours after the first dose of study drug

#### 7 OVERALL DESIGN

This is a Phase 2, randomized, double-blind, placebo-controlled, dose-ranging, 5-arm, parallel study design evaluating the efficacy and safety of VX-548 doses in treating acute pain after a bunionectomy (Figure 7-1).

On Day -1, subjects will undergo a primary unilateral bunionectomy with distal first metatarsal osteotomy (i.e., Austin procedure) and internal fixation under regional anesthesia (Mayo and popliteal sciatic block). A continuous popliteal sciatic block infusion (0.2% ropivacaine) will be started after surgery and remain in place until approximately 3AM, but no later than 5AM, on Day 1. After removal of the popliteal sciatic block, a subject will be randomized to 1 of 5 treatment groups if (1) the subject requests the first dose of study drug for pain relief, (2) the subject's pain is moderate or severe on the VRS, and (3) the subject's pain is ≥4 on the NPRS. If a subject does not meet the VRS and NPRS criteria within 9 hours of removal of the popliteal sciatic block, the subject will not be eligible for this study.

Approximately 202 subjects will be randomized 2:2:1:2:2 to 5 treatment groups: VX-548 (high dose); VX-548 (mid dose); VX-548 (low dose); HB/APAP (opioid reference); or placebo (Table 7-1). Randomization will be stratified by site and baseline NPRS (<8 versus ≥8). To maintain the blind, all subjects will receive the same number of tablets and/or capsules every 6 hours (q6h) in a double-dummy design.

Figure 7-1 VX21-548-101 Study Design



Treatment Period

CRU: clinical research unit; HB/APAP: hydrocodone bitartrate/acetaminophen; NPRS: Numeric Pain Rating Scale; q6h: every 6 hours; VRS: Verbal Categorical Rating Scale

Notes: After removal of the popliteal sciatic block, a subject will be randomized to 1 of 5 treatment groups if (1) the subject requests the first dose of study drug for pain relief, (2) the subject's pain is moderate or severe on the VRS, and (3) the subject's pain is ≥4 on the NPRS. If a subject does not meet the VRS and NPRS criteria within 9 hours of removal of the popliteal sciatic block, the subject will not be eligible for this study.

Table 7-1 VX21-548-101 Treatment Groups

| Treatment | Active Dose | Number of Subjects |
|--------------------|------------------------------------|--------------------|
| VX-548 (high dose) | 100 mg first dose, then 50 mg q12h | 54 |
| VX-548 (mid dose) | 60 mg first dose, then 30 mg q12h | 54 |
| VX-548 (low dose) | 20 mg first dose, then 10 mg q12h | 27 |
| HB/APAP | 5 mg/325 mg q6h | 54 |
| Placebo | | 54 |

HB/APAP: hydrocodone bitartrate/acetaminophen; q6h: every 6 hours; q12h: every 12 hours

Note: To maintain the blind, all subjects will receive the same number of tablets and/or capsules q6h in a double-dummy design. VX-548 active and/or VX-548 placebo will be administered to all subjects q12h: 0 hours (first dose) and at 12, 24 and 36 hours after the first dose of study drug. HB/APAP active or HB/APAP placebo will be administered to all subjects q6h: 0 hours (first dose) and at 6, 12, 18, 24, 30, 36 and 42 hours after the first dose of study drug.

Subjects will report their pain on the NPRS at each scheduled time point through 48 hours after the first dose of study drug. In addition, pain intensity will be recorded on the NPRS immediately before each administration of rescue medication.

Ibuprofen (400 mg orally q6h as needed) will be permitted as a rescue medication for pain relief upon the subject's request starting any time after the first dose of study drug through 48 hours after the first dose of study drug. Subjects are encouraged to wait 90 minutes after the first dose of study drug to receive rescue medication, and subjects should generally not receive rescue medication unless their NPRS is ≥4.

## 7.1 Sample Size and Power

The sample size calculation is based on the comparison between VX-548 and placebo. The primary efficacy endpoint is the time-weighted SPID48 after the first dose. Assuming a standardized effect size of 0.8 for VX-548 (high or mid-dose) compared to placebo as well as a 2-sided significance level of 0.05, 48 evaluable subjects per group would provide at least 90% power. This sample size would allow a minimal detectable standardized effect size of 0.4 to achieve statistical significance between VX-548 (high or mid-dose) and placebo.

Assuming an observed standardized effect size of 0.8, this sample size would provide sufficient precision, with 90% probability for the true standardized effect size greater than 0.53. To allow for withdrawal of up to 10% of randomized subjects over 48 hours of treatment, the study will enroll and randomize approximately 243 subjects in total.

#### 7.2 Randomization

Refer to Section 9.2 of the CSP for details.

#### 7.3 Blinding and Unblinding

Refer to Section 10.7 of the CSP for details.

#### 8 ANALYSIS SETS

#### 8.1 All Subjects Set

The **All Subjects Set** is defined as all subjects who have been randomized or have received at least 1 dose of study drug. This analysis set will be used in subject listings and disposition summary table, unless otherwise specified.

#### 8.2 Full Analysis Set

The **Full Analysis Set (FAS)** is defined as all randomized subjects who have received at least 1 dose of study drug. The FAS will be used to summarize subject demographics, baseline characteristics, and for all efficacy analyses in which subjects will be analyzed according to their randomized treatment group, unless otherwise specified.

#### 8.3 Safety Set

The **Safety Set** is defined as all subjects who have received at least 1 dose of study drug. The Safety Set will be used for all safety analyses in which subjects will be analyzed according to the treatment they received, unless otherwise specified.

#### 9 STATISTICAL ANALYSIS

#### 9.1 General Considerations

The Schedule of Assessments is provided in Section 3 of CSP. The precision standards for reporting variables are provided in an internal Biometrics document that specifies the programming rules including the precision for derived variables.

All individual subject data for subjects who were randomized or received at least 1 dose of study drug will be presented in individual subject data listings.

Continuous variables will be summarized using the following descriptive summary statistics: the number of subjects (n), mean, standard deviation (SD), median, minimum value (min), and maximum value (max), unless otherwise specified.

Categorical variables will be summarized using counts and percentages.

**Baseline value** will be defined as the most recent non-missing measurement (scheduled or unscheduled) collected before the first dose of study drug, unless otherwise specified.

**Change (absolute change) from baseline** will be calculated as post-baseline value – baseline value.

**Treatment-emergent (TE) Period** will include the time from the first dose of study drug in the Treatment Period to either (1) the Safety Follow-up, or (2) the date of the last dose +16 days for subjects who do not have a Safety Follow-up.

**Unscheduled visits:** Unscheduled visit measurements will be included in analysis as follows:

- In scheduled visit windows per specified visit windowing rules
- In the derivation of baseline
- In the derivation of maximum and minimum values during TE period, and maximum and minimum change from baseline values during TE period for safety analyses
- In individual subject data listings as appropriate

**Visit windowing rules:** The analysis visit windows for protocol-defined visits are provided in Appendix A.

**Incomplete/missing data:** For NPRS measurements, missing data will be imputed by applying linear interpolation to the valid observations immediately before and after the missing observation(s). If there are no valid observations after the missing observation(s), the last observation carried forward (LOCF) principle will be applied as a primary approach. Additional details on how to handle missing data is described in subsequent sections when applicable.

**Outliers:** No formal statistical analyses will be performed to detect and/or remedy the presence of statistical outliers, unless otherwise specified.

**Multiplicity:** No multiplicity adjustment will be performed for hypothesis testing. All *P* values for pairwise comparisons in primary efficacy variable, secondary analyses, and other analyses are nominal.

#### 9.2 Background Characteristics

#### 9.2.1 Subject Disposition

The disposition summary will be provided by treatment and overall.

The number of subjects in the following categories will be summarized:

- All Subjects Set
- Randomized
- Full Analysis Set (FAS)
- Safety Set

The number and percentage (based on FAS) of subjects in each of the following disposition categories will be summarized:

• Completed treatment

- Prematurely discontinued treatment and the reason for discontinuation from treatment
- Completed study
- Prematurely discontinued the study and the reason for discontinuation from study

A listing will be provided for subjects who discontinued treatment or who discontinued study with reasons for discontinuation. A randomization listing of subjects will be provided.

#### 9.2.2 Demographics and Baseline Characteristics

Demographics and baseline characteristics will be summarized based on the FAS by treatment group and overall.

Demographic data will include the following:

- Age (in years)
- Sex (male, female)
- Ethnicity (Hispanic or Latino, not Hispanic or Latino, and not collected per local regulations)
- Race (White, Black or African American, Asian, American Indian or Alaska Native, Native Hawaiian or Other Pacific Islander, not collected per local regulations, Other and Multiracial [if 2 or more races reported from a subject])

Baseline characteristics will include the following:

- Weight (kg)
- Height (cm)
- BMI  $(kg/m^2)$
- BMI category ( $<18.5, \ge 18.5 <25, \ge 25 <30, \ge 30 \text{ kg/m}^2$ )
- Site (005, 016, 017, 018, 057, 058, 062, 063)
- NPRS
- NPRS category ( $<8, \ge8$ )
- VRS (moderate, severe)

In addition, data listings will also be provided for:

- Informed consent
- Inclusion/exclusion criteria violation for subjects with any such violations

### 9.2.3 Medical History

Medical history will be coded by using the Medical Dictionary for Regulatory Activities (MedDRA). Medical history will be summarized descriptively based on the FAS by MedDRA system organ class (SOC) and preferred term (PT). This summary will be provided by treatment group and overall. The corresponding data listing will also be provided.

#### 9.2.4 Prior and Concomitant Medications

Medications will be coded using the World Health Organization Drug Dictionary and categorized as the following for the purpose of analysis:

**Prior medication:** Medication that started before the first dose of study drug, regardless of when dosing of the medication ended

**Concomitant medication:** Medication continued or newly received on or after the date of the first dose of study through the end of the TE Period

A given medication may be classified as a prior medication, a concomitant medication, or both a prior and a concomitant medication.

If a medication start date is on or after the first dose date of study drug, then the medication will be classified as a concomitant medication regardless of whether the medication end date is missing or not. If a medication end date is before the first dose date of study drug, then the medication will be classified as a prior medication regardless of whether the medication start date is missing or not.

Note that a medication that started before the first dose of study drug and continued after the first dose will be classified as a prior medication and separately as a concomitant medication. If a medication has a missing or partially missing start/end date and it cannot be determined whether it was taken before the first dose of study drug, or concomitantly, it will be classified as a prior and a concomitant medication.

Details for imputing missing or partial start/stop date and time of medication are described in Appendix B.

Prior and Concomitant medications will be summarized based on the FAS by Preferred Name and listed. This summary will be provided by treatment group and overall.

Supplemental analgesic medications administered after surgery and before removal of the popliteal sciatic block will be included in the Prior medications summary but will be listed separately. Rescue medication will also be included in the summary of Prior medications but will be listed separately.

Prior and concomitant non-pharmacological treatments or procedures will be listed.

## 9.2.5 Study Drug Exposure and Study Drug Compliance

Study drug will be administered to the subjects by site personnel at time points specified in the CSP (Table 3-2 and Section 9.6) during a period of 42 hours. Therefore, it is not needed to perform a calculation of exposure to study drug or a calculation of compliance. All data collected during dispensation of study drug (i.e. time of administration and number of capsules taken) will be presented in an individual data listing only.

## 9.2.6 Important Protocol Deviations

An important protocol deviation (IPD) is a deviation that may significantly affect the completeness, accuracy, or reliability of the study data or that may significantly affect a subject's rights, safety, or well-being. IPD rules will be developed and finalized before

database lock. IPDs will be identified by the PD review team according to the protocol deviation plan.

IPDs will be summarized descriptively by treatment group and overall.

## 9.3 Efficacy Analysis

All efficacy analyses described in this section will be based on the FAS, unless specified otherwise. Subjects will be analyzed according to their randomized treatment assignment. Although the results from the efficacy analyses will be presented as separate pairwise comparisons (i.e. VX-548 versus placebo and HB/APAP versus placebo), all treatment groups will be included in the statistical models described in this section.

#### 9.3.1 Analysis of Primary Endpoint

#### 9.3.1.1 Definition of Primary Endpoint

The primary endpoint is the time-weighted SPID48 after the first dose of study drug. In general, SPID is calculated as:  $\sum \Delta time_i \times PID_i$  where:

- $\Delta \text{time}_i = \text{time}$  (in hours) elapsed since previous measurements
- PID<sub>i</sub> = pain intensity (NPRS) at baseline pain intensity (NPRS) at hour i

Hence:

• SPID48 =  $0.5 \times PID_{0.5} + 0.5 \times PID_1 + 0.5 \times PID_{1.5} + 0.5 \times PID_2 + PID_3 + PID_4 + PID_5 + PID_6 + 2 \times PID_8 + 4 \times PID_{12} + 4 \times PID_{16} + 4 \times PID_{20} + 4 \times PID_{24} + 4 \times PID_{28} + 4 \times PID_{32} + 4 \times PID_{36} + 4 \times PID_{40} + 4 \times PID_{44} + 4 \times PID_{48}$ 

## 9.3.1.2 Primary Analysis

The primary efficacy analysis will be based on an analysis of covariance (ANCOVA) model. The model will include the SPID48 as the dependent variable and treatment as a fixed effect, with site and baseline NPRS as covariates. Data from all treatment groups will be included in the model. If the model estimation does not converge, then site will be removed from the model. The primary results obtained from the model will be the estimated mean treatment effect between VX-548 versus placebo. The Least Squares (LS) mean of the treatment difference for each dose group of VX-548 versus placebo will be provided along with the 95% CI and 2-sided *P* value. In addition, the LS mean with 95% confidence interval (CI) will be provided for each treatment group.

The following imputation scheme will be applied for the primary analysis:

- 1) NPRS scores during the rescue period (within 6 hours after rescue medication) will be replaced by the pre-rescue NPRS.
  - The pre-rescue NPRS will be the NPRS collected immediately before the
    administration of rescue medication, or the last observed NPRS if that score is
    missing. The last observed NPRS can be a score from a regularly scheduled
    measurement or the previous pre-rescue NPRS but cannot be any observed
    scores during the previous rescue period.

- If there are multiple administrations of rescue medication within the same 6-hour period, a local highest NPRS will be used for the imputation during the second 6-hour rescue period. The local highest NPRS is the highest value among the first pre-rescue, the second pre-rescue, and the actual observed (if any) in the overlapping period.
- 2) Missing NPRS scores following treatment discontinuation will be imputed with the last observed or previously imputed NPRS score prior to discontinuation.
- 3) Missing NPRS scores for subjects who completed the treatment but with missing data from certain time point to 48 hours will be imputed with the last observed or previously imputed NPRS score.
- 4) Intermittently missing NPRS scores will be imputed using linear interpolation.

## 9.3.1.3 Supportive Analyses

A supportive analysis based on the Linear trend test will be performed to assess the dose-response relationship. The linear trend test will be based on the LS means obtained from the ANCOVA model from the primary analysis. The 2-sided *P* value will be provided.

#### 9.3.1.4 Additional Analyses

This additional analysis will be performed by modifying the primary analysis in such a way that NPRS scores during the rescue period (within 6 hours after rescue medication) will not be replaced by the pre-rescue NPRS score. The observed NPRS scores will be used instead. The same ANCOVA model as described in Section 9.3.1.2 will be performed.

## 9.3.1.5 Sensitivity Analyses

This sensitivity analysis will be performed by modifying the primary analysis in such a way that missing NPRS scores following treatment discontinuation due to AE will be imputed with the baseline NPRS while the NPRS following treatment discontinuation due to other reasons will be imputed by the last observed or previously imputed NPRS score prior to discontinuation. The same ANCOVA model as described in Section 9.3.1.2 will be performed.

#### 9.3.1.6 Subgroup Analysis

No subgroup analysis for the primary efficacy variable is planned.

For the primary analysis, additional analysis, and sensitivity analysis, SPID48 will also be summarized descriptively, including standard error (SE), by treatment. In addition, NPRS measurements will be summarized descriptively, including SE, by treatment at each scheduled time point and the mean values over time by treatment will be presented in a figure.

## 9.3.2 Analysis of Secondary Efficacy Variables

# 9.3.2.1 Definition of Secondary Efficacy Variables

<u>Time-weighted SPID24 after the first dose of study drug</u>: In general, SPID24 is calculated using the following formula:

• SPID24 =  $0.5 \times \text{PID}_{0.5} + 0.5 \times \text{PID}_1 + 0.5 \times \text{PID}_{1.5} + 0.5 \times \text{PID}_2 + \text{PID}_3 + \text{PID}_4 + \text{PID}_5 + 2 \times \text{PID}_8 + 4 \times \text{PID}_{12} + 4 \times \text{PID}_{16} + 4 \times \text{PID}_{20} + 4 \times \text{PID}_{24}$ 

<u>Proportions of subjects with  $\geq 30\%$ ,  $\geq 50\%$ , and  $\geq 70\%$  reduction in NPRS at 48 hours after the first dose of study drug:</u> Subjects with  $\geq 30\%$ ,  $\geq 50\%$ , and  $\geq 70\%$  reduction in NPRS at 48 hours after the first dose of study drug will be defined as "responders. The percentage reduction in the NPRS will be calculated as following:

• 100% × (NPRS at baseline –NPRS at 48 hours) / NPRS at baseline

The same imputation strategies as described in Section 9.3.1.2 will be applied. However, Subjects who discontinue study drug treatment for any reason prior to 48 hours will be defined as "non-responders" for any of the 3 criteria.

#### 9.3.2.2 Secondary Analyses

<u>Time-weighted SPID24 after the first dose of study drug</u>: SPID24 will be analyzed in the same way as described in Section 9.3.1.2. SPID24 will also be analyzed in the same way as described for SPID48 in Sections 9.3.1.4 and 9.3.1.5.

Proportions of subjects with  $\geq 30\%$ ,  $\geq 50\%$ , and  $\geq 70\%$  reduction in NPRS at 48 hours after the first dose of study drug: Analysis of responder rates at 48 hours between VX-548 and placebo will be conducted using Cochran-Mantel-Haenszel test, stratified by baseline NPRS ( $<8, \geq 8$ ).

#### 9.3.3 Analysis of Other Efficacy Variables

#### 9.3.3.1 Definition of Other Efficacy Variables

Time to onset of "confirmed perceptible pain relief" and "meaningful pain relief" after the first dose of study drug: Time to onset of "first perceptible pain relief" is the time elapsed from first dose of study drug until the subject stops the "first perceptible pain relief" stopwatch. Time to onset of "meaningful pain relief" is the time elapsed from first dose of study drug until the subject stops the "meaningful pain relief" stopwatch. Time to onset of "confirmed perceptible pain relief" will be defined as the time to onset of first perceptible pain relief for those subjects who achieved meaningful pain relief.

If the subject has not stopped the stopwatch by 6 hours after the first dose or the subject receives rescue medication during the first 6 hours, the stopwatch will be stopped and time to onset will be considered censored at 6 hours. If the "first perceptible pain relief" is obtained without subsequent "meaningful pain relief", time to onset of "confirmed perceptible pain relief" will also be considered censored at 6 hours.

Proportions of subjects with  $\geq 30\%$ ,  $\geq 50\%$ , and  $\geq 70\%$  reduction in NPRS at 24 hours after the first dose of study drug: Subjects with  $\geq 30\%$ ,  $\geq 50\%$ , and  $\geq 70\%$  reduction in NPRS at 24 hours after the first dose of study drug will be defined as "responders". The percentage reduction in the NPRS will be calculated as following:

• 100% × (NPRS at baseline –NPRS at 24 hours) / NPRS at baseline

The same imputation strategies as described in Section 9.3.1.2 will be applied. However, Subjects who discontinue the study drug treatment for any reason prior to 24 hours will be "non-responders" for any of the three criteria.

Patient Global Assessment (PGA) of study drug at 48 hours after the first dose of study drug: The PGA of study drug is a single-item assessment of patient perceptions of the method of pain control with the study drug and is evaluated on a 4-point Likert scale (poor, fair, good, or excellent). Subjects with missing PGA at 48 hours will be analyzed as part of a "missing" category.

#### 9.3.3.2 Other Analyses

Time to onset of "confirmed perceptible pain relief" and "meaningful pain relief" after the first dose of study drug: Time to onset of "confirmed perceptible pain relief" will be analyzed using Cox regression model. The model will include treatment as a fixed effect and baseline NPRS as a covariate. Pairwise comparison between VX-548 and placebo will be conducted under the model.

Note: If the placebo group has fewer than 5 subjects experience "confirmed perceptible pain relief", the Cox regression will not be performed. If any other dose group has fewer than 5 subjects experience "confirmed perceptible pain relief", the particular dose group will not be included in the Cox regression model.

Additionally, Kaplan-Meier method will be used to estimate the median time to onset of "confirmed perceptible pain relief" and the survival curve for each treatment group. Logrank test will be used to compare curves between VX-548 and placebo.

Time to onset of "meaningful pain relief" and time to onset of "first perceptible pain relief" will be analyzed in the same way as described for time to onset of "confirmed perceptible pain relief".

Proportions of subjects with  $\geq 30\%$ ,  $\geq 50\%$ , and  $\geq 70\%$  reduction in NPRS at 24 hours after the first dose of study drug: This variable will be analyzed in the same way as described in Section 9.3.2.2 for NPRS responder rates at 48 hours.

Patient Global Assessment (PGA) of study drug at 48 hours after the first dose of study drug: This variable will be summarized descriptively. Cochran-Mantel-Haenszel test, stratified by baseline NPRS ( $\leq$ 8,  $\geq$ 8), will be conducted to compare VX-548 and placebo.

Percentage of subjects using rescue medication, and total rescue medication usage, 0 to 48 hours after the first dose of study drug: The percentage of subjects using rescue medication during 0-48 hours will be analyzed using Cochran-Mantel-Haenszel test, stratified by baseline NPRS ( $<8, \ge 8$ ), to compare VX-548 and placebo. Total rescue medication usage from 0 to 48 hours will be summarized descriptively and Wilcoxon rank-sum test, stratified by baseline NPRS ( $<8, \ge 8$ ), will be conducted to compare VX-548 and placebo.

All analyses described in Sections 9.3.1, 9.3.2 and 9.3.3 on comparisons between VX-548 and placebo will be repeated based on a comparison between HB/APAP and placebo.

## 9.4 Safety Analysis

The overall safety profile of VX-548 will be assessed in terms of the following safety and tolerability endpoints:

- Incidence of treatment-emergent adverse events (TEAEs)
- Clinical laboratory values (hematology, serum chemistry, coagulation studies, and urinalysis)
- ECG outcomes
- Vital signs

All safety analyses will be performed based on the Safety Set by treatment. Only descriptive analyses of safety will be performed, and no statistical hypothesis testing will be performed.

In an unexpected scenario that a subject may receive more than one treatment in the study, the following algorithm will be used to define subject's actual treatment: for any dosed subjects, the actual treatment is defined as the highest dose level among all received VX-548 treatment if the subject received any VX-548 treatment, regardless of the randomized treatment assignment; the actual treatment is defined as HB/APAP if the subject did not receive any VX-548 treatment but did receive any HB/APAP; the actual treatment is defined as placebo only if the subject received placebo at all visits in the study.

#### 9.4.1 Adverse Events

AEs will be coded according to MedDRA. For analysis purposes, AEs will be classified as pretreatment AEs and TEAEs as follows:

**Pretreatment AEs:** AEs that occurred before the first dose of study drug

**Treatment-emergent AEs**: AEs that worsened or started on or after the first dose date of study drug through the end of the TE Period

For AEs with completely missing or partial start dates, if there is no clear evidence that the AEs started before or after the first dose of study drug, the AEs will be classified as TEAEs.

Imputation rules for missing or partial AE start date are defined as Appendix C.

AE summary tables will be presented only for TEAEs, and will include the following:

- All TEAEs
- TEAEs by strongest relationship
- TEAEs by maximum severity
- TEAEs leading to treatment discontinuation
- TEAEs leading to treatment interruption
- Related TEAEs
- Serious TEAEs
- Related serious TEAEs

#### • TEAEs leading to death

Summaries will be presented by MedDRA SOC and PT using frequency counts and percentages (i.e., number and percentage of subjects with an event). When summarizing the number and percentage of subjects with an event, subjects with multiple occurrences of the same AE or a continuing AE will be counted once, and only the maximum severity level will be presented in the severity summaries, and the strongest relationship level in the relationship summaries.

All AEs, including pretreatment AEs and TEAEs will be presented in an individual subject data listing based on the All Subjects Set. In addition, a listing containing individual subject adverse event data for TEAEs leading to treatment discontinuation, TEAEs leading to treatment interruption, SAEs and all deaths will be provided separately.

#### 9.4.2 Clinical Laboratory Assessments

All statistical analyses of laboratory values will be performed using SI units. For treatmentemergent laboratory measurements, the observed values and change from baseline values of the continuous hematology, chemistry, and coagulation results will be summarized at each visit.

The number and percentage of subjects with selected test values meeting threshold analysis criterion event during the TE period will be summarized. The threshold analysis criterion shift from baseline will also be summarized for chemistry measurements. The threshold analysis criteria are provided in Appendix D.

Results of urinalysis and the urine/serum pregnancy test will be in individual subject data listings only.

In addition, a listing of individual subject hematology, chemistry, and coagulation values outside the normal reference ranges will be provided. This listing will include data from both scheduled and unscheduled visits.

## 9.4.3 Electrocardiogram

For the treatment-emergent ECG measurements, a summary of observed values and change from baseline values will be provided at each visit and time point, as applicable, for the following ECG measurements (in msec): heart rate (HR; beats per minute [bpm]), PR interval (msec), RR interval (msec), QRS duration (msec), QT interval (msec), and QT corrected for HR intervals (QTcF [msec]). In addition, the number and percentage of subjects by maximum treatment-emergent value of QT/QTcF intervals, categorized as ≤450 msec, >450 msec and ≤480 msec, >480 msec and ≤500 msec, and >500 msec, as well as maximum treatment-emergent change from baseline value of QT/QTcF intervals, categorized ≤0 msec, and >0 and ≤30 msec, >30 and ≤60 msec, and >60 msec, will be provided.

The number and percentage of subjects meeting threshold analysis criterion during the TE period will be summarized. The threshold analysis criteria are provided Appendix D. A listing containing individual subject measurements meeting the threshold value criteria at any time point will be provided. This listing will include data from both scheduled and unscheduled visits.

#### 9.4.4 Vital Signs

For the treatment-emergent vital signs measurements, the observed values and change from baseline values will be summarized at each visit. The following vital signs parameters will be summarized: systolic and diastolic blood pressure (mm Hg), pulse rate (beats per minute), body temperature (°C), respiratory rate (breaths per minute), oxygen saturation (%).

The number and percentage of subjects meeting threshold analysis criterion during the TE Period will be summarized. The threshold analysis criteria are provided in Appendix D.

In addition, a listing containing individual subject vital signs values will be provided. This listing will include data from both scheduled and unscheduled visits.

## 9.4.5 Physical Examination

Physical examination (PE) results will be presented in individual subject data listings only.

#### 10 SUMMARY OF INTERIM AND IDMC ANALYSES

Not applicable.

#### 11 REFERENCES

Not applicable.

## 12 LIST OF APPENDICES

# Appendix A: Analysis Visit Windows for Safety and Efficacy Assessments

| Assessment | Visit/Time Point <sup>1</sup> | Target Study Day<br>/Time Point per<br>the protocol | Analysis Visit Window<br>(in study days/ time points)<br>2,3,4,5 |
|---|---|---|---|
| Safety Assessment | | | |
| Hematology | Baseline | Day 1 | ≤ Day 1 Pre-dose |
| Serum Chemistry<br>Coagulation | 48 hours | 48 hours | Nominal Visit |
| Standard 12-Lead ECG | Baseline | Day 1 | ≤ Day 1 Pre-dose |
| | 4 hours | 4 hours | Nominal visit for all visits |
| | 16 hours | 16 hours | |
| | 28 hours | 28 hours | |
| | 40 hours | 40 hours | |
| Vital Sign | Baseline | Day 1 | ≤ Day 1 Pre-dose |
| | 2 hours | 2 hours | Nominal visit for all visits |
| | 4 hours | 4 hours | |
| | 24 hours | 24 hours | |
| | 48 hours | 48 hours | |
| | Safety Follow-up | Not applicable | |
| Efficacy Assessment | | | |
| NPRS | Baseline | Day 1 | ≤ Day 1 Pre-dose |
| | At 0.5, 1, 1.5, 2, 3, 4, 5, 6, 8, 12, 16, 20, 24, 28, 32, 36, 40, 44, and 48 hours | At 0.5, 1, 1.5, 2, 3, 4, 5, 6, 8, 12, 16, 20, 24, 28, 32, 36, 40, 44, and 48 hours | ± 5 minutes for 0.5 to 48 hours |
| VRS | Baseline | Day 1 | ≤ Day 1 Pre-dose |
| Rescue Medication | N/A | N/A | [Day 1 post-dose, 48 hours post-dose] |

#### Notes:

- a. If no numerical measurement is available within a visit window, the measurement will be considered missing for the visit.
- b. If there is more than 1 numerical measurement available within the same visit window, use the following rules:

<sup>&</sup>lt;sup>1</sup>Visit/Time point name for analysis purpose is used to report data in tables and figures.

<sup>&</sup>lt;sup>2</sup>The analysis visit windows will be applied using the following rules for both scheduled and unscheduled visits:

- i. The measurement closest to the target day/time point will be used; or
- ii. If there are multiple measurements within the same distance from the target day/time point, the latest measurement will be used.
- iii. If a scheduled and unscheduled measurement have the same date/time, the unscheduled measurement will be used.

<sup>3</sup>For measurements collected on the date of first dose of study drug in Treatment Period, if it cannot be determined whether the measurement is before or after the first dose:

- a. If a scheduled measurement is pre-dose in the CSP, it will be treated as a pre-dose observation. If a scheduled measurement is post-dose in the CSP, it will be treated as a post-dose observation.
- b. Unscheduled measurement will be treated as post-dose observation.

<sup>&</sup>lt;sup>4</sup>When define baseline for efficacy and safety, refer to the generic baseline definition in Section 9.1.

## Appendix B: Imputation Rules for Missing Prior/Concomitant Medication Date

Imputation rules for missing or partial medication start/stop dates are defined below:

- 1. Missing or partial medication start date and time:
  - a. If Hour and/or Minute are missing, do not impute.
  - b. If DAY is missing, use the first day of the month.
  - c. If DAY and Month are both missing, use the first day of the year.
  - d. If DAY, Month and Year are all missing, use a date before the first dose date.
- 2. Missing or partial medication stop date:
  - a. If only DAY is missing, use the last day of the month.
  - b. If DAY and Month are both missing, use the last day of the year.
  - c. If DAY, Month and year are all missing, assign 'continuing' status to stop date.

With missing or partial medication start time, only use the imputed start date to categorize the prior and/or concomitant medication as described in Table 12-2. If hour and/or minute of first dose time are missing, only use the first dose date to categorize the prior and/or concomitant medication. Imputation of missing and/or partial dates for non-pharmacological treatments/procedures will follow the same imputation rule.

Table 12-2 Prior and/or Concomitant Categorization of a Medication

| | <b>Medication Stop Date</b> | |
|---|---|---|
| | < First Dose Date of Study | ≥ First Dose Date and ≤ |
| Medication Start Date | Drug | End Date of TE Period |
| < First dose date of study drug | P | PC |
| $\geq$ First dose date and $\leq$ End date of TE period | - | С |

C: Concomitant; P: Prior

#### Appendix C: Imputation Rules for Missing AE Date and Time

Imputation rules for missing or partial AE start date and time are defined below:

#### If Hour and/or Minute of AE start time are missing, do not impute:

- If the AE start date is before the first dose date, the AE will be classified as pretreatment AE.
- If the AE start date is on or after the first dose date, the AE will be classified as TEAE.

#### If Day of AE start date is missing:

- If the full (or partial) AE end date is NOT before the first dose date or AE end date is missing, then
  - o if the AE start year and month are equal to the month and year of first dose date, then impute the AE start day as the day of first dose date;
  - o else impute the AE start day as 1.
- Else impute the AE start day as 1.

Compare the imputed AE start date with TE period to determine whether the AE is pretreatment AE, or TEAE.

#### If Day and Month of AE start date are missing:

- If the full (or partial) AE end date is NOT before the first dose date or AE end date is missing,
  - o if AE start year is equal to the year of the first dose date, then impute the AE start month and day as the month and day of first dose date.
  - o else impute the AE start Month as January and the Day as 1.
- Else impute the AE start MONTH as January and the DAY as 1.

Compare the imputed AE start date with TE period to determine whether the AE is pretreatment AE, or TEAE.

#### If Year of AE start date is missing:

If the year of AE start is missing or AE start date is completely missing then query site with no imputation. Also compare the full (or partial) AE end date to the first dose date. If the AE end date is before the first dose date then the AE should be considered as a pretreatment AE. Otherwise, the AE will be considered as TEAE.

#### If hour and/or minute of first dose time are missing:

- If the AE start date is before the first dose date, the AE will be classified as pretreatment AE.
- If the AE start date is on or after the first dose date, the AE will be classified as TEAE.

# **Appendix D: Threshold Value Criteria**

Table 12-1 Threshold Analysis Criteria for Laboratory Tests (as applicable)

| Parameter | Threshold Analysis | Comments |
|---|---|---|
| <b>Clinical Chemistry</b> | | |
| ALT | >ULN - ≤3xULN<br>>3x - ≤5xULN<br>>5x - ≤8xULN<br>>8x - ≤20.0xULN<br>>20.0xULN | FDA DILI Guidance Jul 2009. |
| AST | >ULN - ≤3xULN<br>>3x - ≤5xULN<br>>5x - ≤8xULN<br>>8x - ≤20.0xULN<br>>20.0xULN | FDA DILI Guidance Jul 2009. |
| ALT or AST | (ALT>ULN - $\leq$ 3xULN) or (AST>ULN $\leq$ 3xULN)<br>(ALT>3x - $\leq$ 5xULN) or (AST>3x - $\leq$ 5xULN)<br>(ALT>5x - $\leq$ 8xULN) or (AST>5x - $\leq$ 8xULN)<br>(ALT>8x - $\leq$ 20xULN) or (AST>8x - $\leq$ 20xULN)<br>ALT>20xULN or AST>20xULN | - FDA DILI Guidance Jul 2009. |
| Alkaline Phosphatase | >ULN - ≤1.5xULN<br>>1.5 - ≤2.5xULN<br>>2.5 - ≤5.0xULN<br>>5.0 - ≤20.0xULN<br>>20.0xULN | FDA DILI Guidance Jul 2009. |
| Total Bilirubin | >ULN - ≤1.5xULN<br>>1.5 - ≤2xULN<br>>2 - ≤3xULN<br>>3 - ≤10xULN<br>>10xULN | FDA DILI Guidance Jul 2009. |
| Direct Bilirubin | >ULN - ≤1.5xULN<br>>1.5 - ≤2xULN<br>>2 - ≤3xULN<br>>3 - ≤10xULN<br>>10xULN | FDA DILI Guidance Jul 2009. |
| ALT and Total Bilirubin | ALT>3xULN and TBILI>2xULN | FDA DILI Guidance Jul 2009. |
| AST and Total Bilirubin | AST>3xULN and TBILI>2xULN | FDA DILI Guidance Jul 2009. |
| (ALT or AST) and Total Bilirubin | (ALT>3xULN or AST>3xULN) and TBILI>2×ULN | FDA DILI Guidance Jul 2009. |

Table 12-1 Threshold Analysis Criteria for Laboratory Tests (as applicable)

| Parameter | Threshold Analysis | Comments |
|---|---|---|
| GGT | >ULN - ≤2.5xULN<br>>2.5 - ≤5.0xULN<br>>5.0 - ≤20.0xULN<br>>20.0xULN | CTCAE grade 1-4 |
| Albumin | <lln -="" g="" l<br="" ≥30="">&lt;30 - ≥20 g/L<br/>&lt;20 g/L</lln> | CTCAE grade 1-3 |
| Creatinine | >ULN - ≤1.5xULN<br>>1.5 - ≤3.0xULN<br>>3.0 - ≤6.0xULN<br>>6.0xULN | CTCAE grades 1-4 |
| Lipase | >ULN - ≤1.5xULN<br>>1.5x - ≤2xULN<br>>2x - ≤5xULN<br>>5xULN | Criteria based upon CTCAE |
| Total protein | <lln<br>&gt;ULN</lln<br> | No CTCAE |
| Creatine kinase | >ULN - ≤2.5xULN<br>>2.5 - ≤5xULN<br>>5 - ≤10xULN<br>>10xULN | CTCAE grades 1-4 |
| Hematology | | |
| Hemoglobin | Hgb decreased (anemia) <lln -="" <100="" <80="" g="" l="" l<="" td="" ≥100="" ≥80=""><td>CTCAE grade 1-3</td></lln> | CTCAE grade 1-3 |
| | Hgb increased >ULN - ≤20 g/L above ULN >20 g/L above ULN - ≤40 g/L above ULN >40 g/L above ULN | CTCAE grade 1-3 |
| Platelets | Platelet decreased <lln -="" 10e9="" <25.0="" <50.0="" <75.0="" l="" l<="" td="" x="" ≥25.0="" ≥50.0="" ≥75.0=""><td>CTCAE grade 1-4</td></lln> | CTCAE grade 1-4 |
| | Platelet increased >ULN | No CTCAE available |
| Coagulation | | |
| Activated partial thromboplastin time (PTT) | >ULN - ≤1.5xULN<br>>1.5 - ≤2.5xULN<br>>2.5xULN | CTCAE grade 1-3 |

Table 12-1 Threshold Analysis Criteria for Laboratory Tests (as applicable)

| Parameter | Threshold Analysis | Comments |
|---|---|---|
| Prothrombin time (PT)<br>International | >ULN - ≤1.5xULN<br>>1.5 - ≤2.5xULN | CTCAE grade 1-3 |
| Normalized Ratio (INR) | >2.5 x ULN | |

Table 12-2 Threshold Analysis Criteria for ECGs

| Parameter | Threshold Analysis | Comments |
|---|---|---|
| HR | Bradycardia <50 bpm <45 bpm Decrease from baseline ≥10 bpm | Per HV grade 2, 3, plus shift change |
| | Decrease from baseline ≥20 bpm <50 bpm and decrease from baseline ≥10 bpm <50 bpm and decrease from baseline ≥20 bpm | |
| | Tachycardia >100 bpm >115 bpm >130 bpm Increase from baseline ≥10 bpm Increase from baseline ≥20 bpm >100 bpm and increase from baseline ≥10 bpm >100 bpm and increase from baseline ≥20 bpm | Per HV grade 1, 2, 3, plus shift change |
| PR | ≥240 ms<br>≥300 ms<br>≥200 ms and increase from baseline ≥40 ms<br>≥200 ms and increase from baseline ≥100 ms | |
| QRS | >110 ms >160 ms Increase from baseline ≥20 ms Increase from baseline ≥40 ms | |
| QTc | >450 to <500ms (Male) or >470 to <500ms (Fem ≥500 ms Increase from baseline Increase from baseline >10 ms Increase from baseline >20 ms Increase from baseline >40 ms Increase from baseline >60 ms | ale) To be applied to any kind of QT correction formula. |

Table 12-3 Threshold Analysis Criteria for Vital Signs

| Parameter | Threshold Analysis | Comments |
|---|---|---|
| Pulse Rate | Same as above in ECG category | |
| SBP increased | >140 mmHg<br>>160 mmHg<br>>10 mmHg increase from baseline | |
| | >20 mmHg increase from baseline | |
| | >140 mmHg & >10 mmHg increase from baseline | |
| | >140 mmHg & >20 mmHg increase from baseline | |
| | >160 mmHg & >10 mmHg increase from baseline<br>>160 mmHg & >20 mmHg increase from baseline | |
| SBP decrease | <90 mmHg | Per HV grade 1, 3, plus shift change |
| | <80 mmHg | |
| | >10 mmHg decrease from baseline<br>>20 mmHg decrease from baseline | |
| | 20 mining decrease from basefine | |
| | <90 mmHg and >10 mmHg decrease from baseline | |
| | <90 mmHg and >20 mmHg decrease from baseline | |
| | <80 mmHg and >10 mmHg decrease from baseline<br><80 mmHg and >20 mmHg decrease from baseline | |
| DBP increased | >90 mmHg | |
| DBI mercused | >100 mmHg | |
| | >5 mmHg increase from baseline | |
| | >10 mmHg increase from baseline | |
| | >90 mmHg and >5 mmHg increase from baseline | |
| | >90 mmHg and >10 mmHg increase from baseline | |
| | >100 mmHg and >5 mmHg increase from baseline | |
| DDD 1 1 | >100 mmHg and >10 mmHg increase from baseline | |
| DBP decreased | <60 mmHg<br><45 mmHg | |
| | >5 mmHg decrease from baseline | |
| | >10 mmHg decrease from baseline | |
| | - | |
| | <60 mmHg and >5 mmHg decrease from baseline | |
| | <60 mmHg and >10 mmHg decrease from baseline | |
| | <45 mmHg and >5 mmHg decrease from baseline<br><45 mmHg and >10 mmHg decrease from baseline | |
| Oxygen saturation | <88% | |
| decreased | <95% and decrease from baseline >5% of absolute oxygen saturation | |